CLINICAL TRIAL: NCT04844112
Title: Assessment of the Real-time CT/MR-US Automatic Fusion System Using Vascular Matching in Pre-procedure Planning for Radiofrequency Ablation: Preliminary Study
Brief Title: CT/MR-US Automatic Fusion System in Pre-procedure Planning for Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1506-015-677
Record Dates: First submitted 2021-04-06; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiofrequency ablation; Fusion imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): patients undergo routine conventional feasibility planning ultrasound, and clinical decision of RFA feasibility is made based on conventional planning ultrasound.
  Then additional planning ultrasound using automatic CT/US fusion technique is immediately performed by the same operator, and clinical decision is made based on fusion imaging.
  Interventions: Procedure: automatic CT/MRI-US fusion system guided radiofrequency ablation

INTERVENTIONS:
Procedure: automatic CT/MRI-US fusion system guided radiofrequency ablation — automatic CT/MRI-US fusion system guided radiofrequency ablation

SUMMARY:
To prospectively evaluate the technical success rate of real-time computed tomography/CT/magnetic resonance imagingMR and -ultrasound (CT/MRI-US) automatic fusion system and the long-term therapeutic efficacy of radiofrequency ablation (RFA) guided by automatic fusion in hepatocellular carcinoma (HCC) patients.

DETAILED DESCRIPTION:
RFA is one of commonly used local therapies for primary or secondary liver tumors. For successful and safe procedure, safe route of electrode and lesion visibility are essential for RFA, and the conditions are usually evaluated on pre-RFA planning ultrasonography (USG). However, RFA is sometimes aborted due to limited sonic window of various cause and challenging identification of small isoechoic tumors or hepatocellular carcinomas among dysplastic nodules . Therefore, precise targeting and assuring safe route would be of clinical importance. In this preliminary study, investigators attempted to determine automatic US and CT/MR fusion technique would be able to improve RFA feasibility in patients with liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or typical imaging based diagnosis of HCC
* Multiphase CT or MRI within 3 months ahead of procedure
* No evidence of distant metastasis
* No contraindications for conventional RFA procedure in our institute, which are uncontrolled coagulopathy (international standard ratio ≥ 1.6, or platelet > 50,000), poor cooperation, unfeasible for sedation, portal vein tumor thrombus, tumor number >4, largest tumor size > 5cm, and tumors abutting portal vein or bile ducts bigger than segmental branches.

Exclusion Criteria:

* Lack of multiphase CT or MRI withing 3 months ahead of procedure
* RFA planned for palliative purpose
* Diagnosed as non-HCC malignancy
* Right hepatectomy state

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Technical success rate of the fusion process | Immediately after fusion process
  Absolute technical success rate of the fusion process
Technical success rate of the overall RFA procedure | immediately after RFA procedure
  Absolute technical success rate of the overall RFA compared to literature
Rate of complete ablation of the tumor after 1 month clinical follow up | 1 month after the RFA procedure
  Rate of complete ablation of the tumor after 1 month clinical follow up compared to literature

SECONDARY OUTCOMES:
Local tumor progression rate | During post procedural follow up to 5 years
  Local tumor progression rate after follow up compared to literature
Tumor visibility before and after the fusion process | 10 minutes after finishing planning USG
  Tumor visibility recorded by a 4-scale scoring system. Comparison between pre- and post- fusion process.
Technical feasibility before and after the fusion process | 10 minutes after finishing planning USG
  Technical feasibility recorded by a 4-scale scoring system. Comparison between pre- and post- fusion process.
Safety of the approach route before and after the fusion process | 10 minutes after finishing planning USG
  Safety of the approach route recorded by a 4-scale scoring system. Comparison between pre- and post- fusion process.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, Study Chair — Professor

IPD SHARING:
Plan to Share IPD: No